CLINICAL TRIAL: NCT02677532
Title: Analgesia Postoperatoria Mediante Catetere Perdurare e Analgesia Postoperatoria Mediante Infusione Continua Periferia Nell'Intervento Chirurgico Per Riparazione Chirurgica di Aneurismi Dell'Aorta Addominale: Tecniche a Confronto
Brief Title: Epidural Versus Wound Infusion Plus Morphine Bolus in Open Abdominal Aortic Aneurysm Repair
Acronym: APERIVIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Paolo Pelosi, Professor, University of Genova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APERIVIP
Record Dates: First submitted 2016-01-29; First posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Morphine; Levobupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural infusion (Active Comparator): Thoracic epidural bolus of 10 ml levobupivacaine 0.25% plus sufentanil 0.15 mcg/kg before end of surgery, followed by continuous epidural infusion of 0.12% levobupivacaine plus 0.4 mcg/ml at 5 ml/h infusion rate for 48 hours.
  Interventions: Drug: Paracetamol; Drug: Levobupivacaine epidural bolus; Drug: Sufentanil epidural bolus; Device: Epidural catheter placement; Drug: Levobupivacaine plus sufentanil epidural infusion
- Wound infusion plus morphine bolus (Experimental): Intravenous slow bolus of 10 mg morphine, wound infiltration with 10 ml levobupivacaine 0.5%, followed by pre-peritoneal continuous wound infusion of levobupivacaine 0.25% at 4 ml/h infusion rate for 48 hours.
  Interventions: Drug: Paracetamol; Drug: Levobupivacaine wound infiltration; Drug: Morphine; Device: Wound infusion catheters placement; Drug: Levobupivacaine wound infusion

INTERVENTIONS:
Drug: Paracetamol — 1 g every 8 hours
Drug: Levobupivacaine wound infiltration — Wound infiltration with 10 ml levobupivacaine 0.5%
  Arms: Wound infusion plus morphine bolus
Drug: Levobupivacaine epidural bolus — Epidural bolus of 10 ml 0.25% levobupivacaine
  Arms: Epidural infusion
Drug: Sufentanil epidural bolus — Epidural bolus of 0.15 mcg/kg sufentanil
  Arms: Epidural infusion
Drug: Morphine — Intravenous slow bolus of 10 mg morphine
  Arms: Wound infusion plus morphine bolus
Device: Epidural catheter placement — Thoracic epidural catheter placement in the T7-T8 or T8-T9 intervertebral space
  Arms: Epidural infusion
Device: Wound infusion catheters placement — Pre-peritoneal placement of two catheters for wound infusion
  Arms: Wound infusion plus morphine bolus
Drug: Levobupivacaine plus sufentanil epidural infusion — Epidural infusion of levobupivacaine 0.12% plus sufentanil 0.4 mcg/ml at 4 ml/h for 48 h
  Arms: Epidural infusion
Drug: Levobupivacaine wound infusion — Wound infusion with levobupivacaine 0.25% at 4 ml/h for 48 h
  Arms: Wound infusion plus morphine bolus

SUMMARY:
The aim of the study is to determine wether continuous wound infusion with local anaesthetic plus a single dose intravenous morphine is non-inferior to postoperative analgesia provided with continuous thoracic epidural infusion of local anaesthetic plus opiate, in patients undergoing open abdominal aortic aneurism repair.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective open aortic aneurism repair

Exclusion Criteria:

* Patient refusal
* Platelet count < 80*10^3/mcL
* International Normalised Ratio > 1.5
* Other contraindications to the placement of epidural catheter, including ongoing anti platelet or anticoagulant treatment not suspended according to national guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Average postoperative pain assessed with numeric rating scale (NRS) in the first 48 hours | Average of the NRS recorded at the different time-points (up to 48 hours after emergence from general anaesthesia)

SECONDARY OUTCOMES:
Need for rescue doses of morphine at each time-point | 0, 4, 8, 12, 24, 36, 48 hours after emergence from general anaesthesia
  Need for a bolus of 5 mg intravenous morphine to relief pain
Number of patients requiring oxygen administration at each time-point | 0, 4, 8, 12, 24, 36, 48 hours after emergence from general anaesthesia
Number of patients that have restored bowel function at each time-point | 0, 4, 8, 12, 24, 36, 48 hours after emergence from general anaesthesia
  Time to first stool analysis
Number of patients whose urinary catheter was removed at each time-point | 0, 4, 8, 12, 24, 36, 48 hours after emergence from general anaesthesia
  Time to catheter removal analysis
Number of patients that have restored ability to walk at each time-point | 0, 4, 8, 12, 24, 36, 48 hours after emergence from general anaesthesia
Non-invasive blood pressure (mmHg) at each time-point | 0, 4, 8, 12, 24, 36, 48 hours after emergence from general anaesthesia
  Blood pressure (systolic, diastolic, mean in mmHg)
Length of hospital stay | Follow-up of up to 3 months after surgery
Heart rate (bpm) at each time-point | 0, 4, 8, 12, 24, 36, 48 hours after emergence from general anaesthesia
Incidence of postoperative nausea and vomiting | 0, 4, 8, 12, 24, 36, 48 hours after emergence from general anaesthesia

OTHER OUTCOMES:
Incidence of postoperative cardiovascular adverse events | Intra-hospital follow-up of up to 3 months after surgery
Incidence of postoperative pulmonary complications | Intra-hospital follow-up of up to 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- UO Anestesia e Terapia Intensiva, IRCCS AOU San-Martino IST, Genova, Genova, Italy

IPD SHARING:
Plan to Share IPD: No